CLINICAL TRIAL: NCT04329078
Title: Relevance of Sensitization to Legumes in Children Allergic to Peanut
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI247
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Allergy;Food
Keywords: food allergy; peanut; legumes; sensitization
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this study are to determine in children allergic to peanut (i) the prevalence of sensitization to other legumes, (ii) the prevalence of allergy to each legume in patients who are sensitized to it (iii ) the severity of the allergy to legumes other than peanut

DETAILED DESCRIPTION:
Allergy to legumes is more and more frequent, especially in children allergic to peanut, with some severe reactions but little is known about cross-reactivity and clinical meanings of legumes sensitization in children allergic to peanut.

All children with a confirmed peanut allergy and followed at the University Hospital of Nancy between January 1st 2017 and February 29th 2020 will be included in order to evaluate the prevalence of sensitization and allergy to other legumes in this population.

In children allergic to peanut and to at least one other legume, we will evaluate the severity of the allergy and the sIgE profiles for peanut.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed allergy to peanut

Exclusion Criteria:

* no available information regarding sensitization and tolerance to legumes

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children allergic to peanut with a follow-up at the Pediatric Allergy Department of the University Hospital of Nancy from january 2017 to february 2020
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
sensitization to legumes | 2017 to 2020
  skin and sIgE sensitization

SECONDARY OUTCOMES:
allergy to legumes | 2017 to 2020
  history of allergic reaction or oral food challenge
severity of allergy to legumes | 2017 to 2020
  history of allergic reaction or oral food challenge

IPD SHARING:
Plan to Share IPD: No